CLINICAL TRIAL: NCT04498871
Title: Managed Access Program (MAP) to Provide Access to Nilotinib, for Patients With Hypereosinophilic Syndrome (HES)
Brief Title: MAP to Provide Access to Nilotinib, for Patients With HES
Status: No longer available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAMN107A2413
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Hypereosinophilic Syndrome (HES)
Keywords: Nilotinib; Hypereosinophilic syndrome; HES
MeSH Terms: conditions — Hypereosinophilic Syndrome | interventions — nilotinib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Nilotinib — Nilotinib is recommended to be administered orally on a continuous schedule at a dose of 400 mg twice daily. The patient should be instructed to take each morning dose of nilotinib 2 hours after a light breakfast (e.g., toast and jam), with no oral intake other than water for 1 hour after dosing. It is recommended that the patient take nilotinib doses every 12 hours with a glass of water. The evening dose of nilotinib should be taken at least 2 hours after dinner with no oral intake other than water for 1 hour after dosing.

SUMMARY:
The purpose of this program is to allow access to nilotinib for eligible patients diagnosed with Hypereosinophilic syndrome (HES). The patient's Treating Physician should follow the suggested treatment guidelines and comply with all local health authority regulations. The requesting Treating Physician submitted a request for access to drug (often referred to as Compassionate Use) to Novartis which was reviewed and approved by the medical team experienced with the drug and indication. Please refer to the latest Investigator's Brochure (IB) or approved label for overview of drug including: non-clinical and clinical experience, risk and benefits. Novartis will continue to provide any new safety information to the Treating Physician as they emerge.

ELIGIBILITY:
Inclusion criteria

1. ≥ 18 years of age
2. Hypereosinophilic syndrome/chronic eosinophilic leukemia who have a clinical indication for treatment and meet the following criteria (Vandenberghe, et al 2004):

   * eosinophilia greater than 1500/mm3 which persists greater than 6 months
   * exclusion of other causes of eosinophilia including clonal or abnormal T-cell populations, exclusion of reactive eosinophilia, and malignancies or T-cell disorders associated with eosinophilia
   * signs and symptoms of organ involvement
3. WHO Performance status of ≤ 2
4. Patient must have the following laboratory values:

   * Potassium ≥ LLN (lower limit of normal) or corrected to within normal limits with supplements prior to the first dose of AMN107
   * Total calcium (corrected for serum albumin) ≥ LLN or correctable with supplements
   * Magnesium ≥ LLN or corrected to within normal limits with supplements prior to the first dose of AMN107
   * Phosphorus ≥ LLN or correctable with supplements
   * ALT and AST ≤ 2.5 x ULN or ≤ 5.0 x ULN if considered due to tumor
   * Alkaline phosphatase ≤ 2.5 x ULN unless considered due to tumor
   * Serum bilirubin ≤ 1.5 x ULN
   * Serum creatinine ≤ 1.5 x ULN
   * Serum amylase ≤ 1.5 x ULN and serum lipase ≤ 1.5 x ULNWritten patient informed consent must be obtained prior to start of treatment.

Written patient informed consent must be obtained prior to start of treatment.

Exclusion criteria

Patients eligible for this Treatment Plan must not meet any of the following criteria:

1. History of hypersensitivity to any drugs or metabolites of similar chemical classes as nilotinib. Any exclusionary sites of disease (e.g., brain metastases).
2. Impaired cardiac function
3. Patients who have undergone major surgery ≤ 2 weeks prior to Visit 1 or who have not recovered from side effects of such surgery
4. Known Cytopathologically confirmed CNS infiltration.
5. Use of therapeutic warfarin.
6. Acute or chronic liver or renal disease considered unrelated to tumor.
7. Treatment with any hematopoietic colony-stimulating growth factors ≤ 1 week prior to starting Nilotinib. Erythropoietin is allowed.
8. Patient who has not recovered from side effects of prior chemotherapy, immunotherapy, other investigational drugs, wide field radiotherapy, or major surgery. Patient who has received imatinib < 5 days prior to AMN107 or has not recovered from side effects of therapy. Hydroxyurea is permitted during the first 28 days of treatment (up to 5 g/day) for a maximum of 7 days.
9. Patient with a history of another primary malignancy that is currently clinically significant or requires active intervention.
10. Known diagnosis of human immunodeficiency virus (HIV).
11. Known ongoing alcohol or drug abuse
12. Unwillingness or inability to comply with the treatment protocol including returning for scheduled visits
13. Participation in a prior investigational study within 30 days prior to enrollment or within 5-half lives of the investigational product, whichever is longer.
14. Pregnant or nursing (lactating) women,

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult